CLINICAL TRIAL: NCT06140238
Title: Preemptive Analgesic Efficacy of Parecoxib for Reducing Postoperative Pain in Gynecological
Brief Title: Preemptive Analgesic Efficacy of Parecoxib for Reducing Postoperative Pain in Gynecological Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 113/2566
Record Dates: First submitted 2023-08-28; First posted 2023-11-18 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2023-08

CONDITIONS: Preemptive Analgesia; Gynecological Surgery; Postoperative Pain; Parecoxib
Keywords: Preemptive analgesia; Gynecological surgery; Parecoxib; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — parecoxib; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Groups of patients who have Parecoxib drug administration before start surgery
  Interventions: Drug: Parecoxib
- Control group (Placebo Comparator): Group of patients who have normal saline (Placebo) administration before start surgery
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Parecoxib — Parecoxib administration 15 minutes before start surgical operation
  Arms: Experimental group
Drug: Normal saline — Normal saline administration 15 minutes before start surgical operation
  Arms: Control group

SUMMARY:
The research is to test the preemptive analgesic efficacy of Parecoxib drug in gynecological surgery by comparing Parecoxib drug and NSS administration 15 min before starting the surgery which the result of postoperative pain score is interpret by visual analog scale index

DETAILED DESCRIPTION:
The research is working on testing the preemptive analgesic efficacy of Parecoxib drug in gynecological surgery whether its can reduce postoperative pain score, reduce total opioid consumption in first 24 hour postoperation and reduce postoperation hospital length stay. Patients who are undergoing gynecological surgery is recruited to the research project while they admit in the hospital for preoperative preparation, in each type of surgery groups (1.Total abdominal hysterectomy 2. Adnexal surgery 3. Surgical staging) will divided in to 2 groups which is experimental group (Parecoxib) and control group (Normal saline). The experimental group will have Parecoxib administration 15 min before starting the surgery and control group will have normal saline administration 15 min before starting the surgery as same, the primary result is postoperative pain score which is interpreted by Visual analog scale index at 2,6,12,24 hour postoperation, the patients will get opioid drug (Morphine) for pain control depending on pain score index they inform, if pain score >7: morphine 0.075 mg/kg iv, if pain score 5 : morphine 0.05mg/kg iv, if pain score <5 : no morphine given. Lastly the side effect of Parecoxib drug will be observed and postoperative hospital length stay of each patient will be recorded

ELIGIBILITY:
Inclusion Criteria:

* Female patients age between 18-70 year-old, who participate in explor lap gynecological surgery (Hysterectomy, Adnexal surgery and surgical stagings) using general anesthesia technique
* American society of Anesthesiologists physical status grade I-II
* Capable to communicate in Thai language

Exclusion Criteria:

* Allergic to NSAIDs and opioid
* Allergic to Parecoxib drug
* Underlying neuropathic pain
* Pregnant woman or woman who undergoes breast feeding
* Uncontrolled hypertension disease, BP >160/110 at admission date
* Underlying ischemic heart disease, Ischemic stroke or peripheral arterial disease
* History status post coronary artery bypass grafting
* Patients who take Aspirin within 7 days before surgery date
* Had underlying which is contraindiated to NSAIDs drug such as Gastritis, history of GI ulcer, chronic kidney disease (Cr clearance < 30ml/min), liver cirrhosis (Child-Pugh class B or above/ serum albumin < 25 g/l)
* Patients who had NSAIDs drug while admit in hospital for preparing the operation before surgery date

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 178 (Actual)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-04-27 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Post operative pain score | 24 hour post operation
  Post operative pain score at 2,6,12,24 hr, described by 'Visual analog pain scale'

SECONDARY OUTCOMES:
Total dose of opioid drug consumption | 24 hour post operation
  Total dose of opioid drug consumption (Morphine) in 24 hour post operation

OTHER OUTCOMES:
Side effect from Parecoxib drug | 24 hour post operation
  observe any side effects of Parecoxib drug which are nausea, vomit and respiratory depression
Total hospital length stay after operation | Post operation date to discharge date
  record total hospital length stay since post operation date to discharge date

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
drafting official document and distribute to IPD about study protocal, statistical analysis plan. inform consent and clinical study report
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 10 September 2023 to 27 June 2024